CLINICAL TRIAL: NCT06793917
Title: Tislelizumab Plus FOLFOX Versus POF in the Treatment of Locally Advanced Unresectable or Metastatic Gastric/Gastroesophageal Junction Adenocarcinoma
Brief Title: Tislelizumab Plus FOLFOX Versus POF in the Treatment of Locally Advanced: a Multicenter, Open-label, Randomized Phase III Studyunresectable or Metastatic Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYLT-030
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab; Oxaliplatin; Levoleucovorin; Fluorouracil; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab combined with POF (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Oxaliplatin injection; Drug: Levo-Leucovorin; Drug: 5-fluorouracil; Drug: Paclitaxel
- Tislelizumab combined with mFOLFOX6 (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Oxaliplatin injection; Drug: Levo-Leucovorin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab will be administered on day 1 of each cycle at 200mg once every 14 days.
Drug: Oxaliplatin injection — Oxaliplatin will be administered on day 1 of each cycle at 85mg/m2 once every 14 days.
Drug: Levo-Leucovorin — Levo-Leucovorin will be administered on day 1 of each cycle at 200 mg/m2 once every 14 days.
Drug: 5-fluorouracil — 5-fluorouracil will be administered at 2400 mg/m2 over 46-hour every 14 days.
Drug: Paclitaxel — Paclitaxel will be administered on day 1 of each cycle at 135mg/m2
  Arms: Tislelizumab combined with POF

SUMMARY:
To compare the efficacy and safety of tislelizumab combined with FOLFOX or combined with POF in the treatment of locally advanced unresectable or metastatic gastric/gastroesophageal junction adenocarcinoma with CPS≥1

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced unresectable, histologically confirmed adenocarcinoma of the gastric or gastroesophageal junction.
* 18-70yeas.
* ECOG PS 0-1.
* No previous chemotherapy (perioperative chemotherapy, six months after fluorouracil alone or one year after oxaliplatin or a combination of taxoid and fluorouracil can be included), radiotherapy or immunotherapy.
* With normal marrow, liver and renal function: a hemoglobin (HGB) of ≥100g/L (without blood transfusion during 14 days); a leucopenia count of ≥4.0×109/L; a platelet count of ≥100×109/L; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault); a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis.
* Life expectancy ≥3 months.
* With normal electrocardiogram results and no history of congestive heart failure.
* With normal coagulation function: activated partial thromboplastin time (APTT), prothrombin time (PT) and INR, each ≤ 1.5 x ULN.
* Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of Tislelizumab until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug.
* With written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.
* Have a known PD-L1 CPS/MMR (or MSI) /HER2(FISH) test result, or have sufficient samples for relevant testing.

Exclusion Criteria:

* Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer.
* Patients with brain or central nervous system metastases, including leptomeningeal disease.
* Pregnant (positive pregnancy test) or breast feeding.
* Serious, non-healing wound, ulcer, or bone fracture.
* Significant cardiac disease as defined as: unstable angina, New York Heart Association (NYHA) grade II or greater, congestive heart failure, history of myocardial infarction within 6 months Evidence of bleeding diathesis or coagulopathy.
* History of a stroke or CVA within 6 months.
* Clinically significant peripheral vascular disease.
* HIV-positive, active hepatitis B or C (HBV, HCV);
* Inability to comply with study and/or follow-up procedures.
* Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.
* Her2-positive (IHC 3+ or 2+/FISH+) patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Estimated)
Dates: Start 2025-06-07 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 4 years
  The length of time from enrollment until the time of progression of disease (PFS, progression-free survival)

SECONDARY OUTCOMES:
Objective response rate | every 4 weeks
  Clinical response of treatment according to RESIST v1.1 criteria (ORR, objective response rate)
Overall survival | 4 years
  The length of time from enrollment until the time of death (OS, overall survival).

CONTACTS AND LOCATIONS:
Overall Officials: Rong bo Lin, bachelor, Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Fujian cancer hospital, Fuzhou, Fujian, China